CLINICAL TRIAL: NCT01708538
Title: Phase III Study of Corneal Collagen Cross-linking Using Two Different Techniques.
Brief Title: The Effects of Corneal Collagen Cross-linking
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rush Eye Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Rush CXL
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Corneal Ectasia Disorders Including Keratoconus
Keywords: keratoconus, corneal collagen crosslinking, riboflavin, corneal ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epithelium on (Active Comparator): Epi not removed during CXL treatment
  Interventions: Drug: CXL
- Epithelium off (Active Comparator): Epi removed before CXL treatment
  Interventions: Drug: CXL

INTERVENTIONS:
Drug: CXL — corneal crosslinking

SUMMARY:
The corneal collagen cross-linking treatment has been used with increasing success to treat corneal dystrophies such as "keratoconus." Recent advances have allowed different techniques for performing this cross-linking treatment. This study investigates the effects of corneal cross-linking using different surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-70, willing to participate, diagnosis of corneal ectasia disorder

Exclusion Criteria:

* Unwilling or unable to participate in trial

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  Best corrected Snellen acuity
Keratometry measurements | 1 year
  Average curvature of the cornea

CONTACTS AND LOCATIONS:
Locations (1):
- Rush Eye Associates, Amarillo, Texas, United States

REFERENCES:
- [Derived] Rush SW, Rush RB. Epithelium-off versus transepithelial corneal collagen crosslinking for progressive corneal ectasia: a randomised and controlled trial. Br J Ophthalmol. 2017 Apr;101(4):503-508. doi: 10.1136/bjophthalmol-2016-308914. Epub 2016 Jul 7. PMID 27388250